CLINICAL TRIAL: NCT00254384
Title: Neoadjuvant Chemotherapy With Docetaxel, Cisplatin Followed by Maintenance Therapy With the EGFR Inhibitor Erlotinib (Tarceva) in Patients With Stage I, II and III Non-Small Cell Lung Cancer Following Definitive Surgical Resection
Brief Title: Docetaxel, Cisplatin, and Erlotinib Hydrochloride in Treating Patients With Stage I-III Non-small Cell Lung Cancer Following Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0221; NCI-2012-01560 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-00817; 2004-0221 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IA Lung Non-Small Cell Carcinoma AJCC v7; Stage IB Lung Non-Small Cell Carcinoma AJCC v7; Stage IIA Lung Non-Small Cell Carcinoma AJCC v7; Stage IIB Lung Non-Small Cell Carcinoma AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (docetaxel, cisplatin, erlotinib hydrochloride) (Experimental): Patients receive docetaxel IV over 1 hour followed by cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning within 90 days following definitive surgical resection, patients receive erlotinib hydrochloride PO daily for up to 1 year.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Erlotinib; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Erlotinib — Given PO
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies docetaxel, cisplatin, and erlotinib hydrochloride in treating patients with stage I-III non-small cell lung cancer following surgery. Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving docetaxel, cisplatin, and erlotinib hydrochloride together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety/toxicity of neoadjuvant chemotherapy with cisplatin and docetaxel followed by maintenance therapy with the epidermal growth factor receptor (EGFR) inhibitor erlotinib (erlotinib hydrochloride) in patients with stage I-III non-small cell lung cancer (NSCLC) undergoing definitive treatment with surgery and/or radiation.

II. To estimate the agreement in baseline to post-treatment changes of EGFR expression (i.e., EGFR modulation) between buccal smears and bronchial tissue.

SECONDARY OBJECTIVES:

I. To evaluate the disease free survival of this therapeutic combination. II. To assess overall quality of life. III. To evaluate predictive biomarkers in early-stage NSCLC.

OUTLINE:

Patients receive docetaxel intravenously (IV) over 1 hour followed by cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning within 90 days following definitive surgical resection, patients receive erlotinib hydrochloride orally (PO) daily for up to 1 year.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of stage I, II or III non-small cell lung cancer; tissue blocks or slides will be requested
* Patients must have surgically resectable disease and may not be treated with prior chemotherapy or radiation
* Patients must be able to tolerate systemic chemotherapy prior to surgical resection
* No acute intercurrent illness or infection
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Leukocytes >= 3,000/uL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 8g/dL
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Bilirubin within normal institutional limits
* Alkaline phosphatase (alk phos) =< 2.5 x upper limit of normal (ULN); if alk phos > 2.5 x ULN but =< 5 x ULN, patient is eligible if AST or ALT =< ULN
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 1.5 x ULN; if AST or ALT > 1.5 x ULN but =< 5 x ULN, patient is eligible if alk phos is =< ULN
* Prior to study enrollment, all women of child-bearing potential must have a negative pregnancy test; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 2 months after the completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with a history of non-melanoma skin cancer, or other malignancies treated 5 years or more prior to the current tumor, from which the patient has remained continually disease-free, are eligible
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior chemotherapy or radiotherapy for lung cancer
* Patients may not be receiving any other investigational agents within 30 days of trial entry, including anti-EGFR drugs
* Patient has signs or symptoms of acute infection requiring systemic therapy
* Patient exhibits confusion, disorientation, or has a history of major psychiatric illness that may impair patient's understanding of the informed consent
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Functional Classification class II or worse), unstable angina pectoris, serious or clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients refusing to sign the informed consent
* Patients with pre-existing peripheral neuropathy National Cancer Institute (NCI) Common Toxicity Criteria (CTC) grade 2 or worse
* Patients must not be pregnant or breast-feeding and all (male and female) must use a contraceptive method deemed acceptable by the investigator while receiving active treatment in the study and for up to two months following completion of therapy
* Patients with a history of severe hypersensitivity reaction to Taxotere and or polysorbate 80 must be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-10-05 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Rate of grade 3 or greater toxicities (hematologic or non-hematologic) | Up to 5 years post-treatment
Changes of EGFR expression (i.e., EGFR modulation) between buccal smears and bronchial tissue | From baseline up to 5 years post-treatment
  Agreement will be estimated using the kappa coefficient. An important aspect of this trial is to identify changes in expression of potential biomarkers between buccal smears and bronchial tissues after induction (neoadjuvant) platinum-based therapy in early-stage , resectable non-small cell lung cancers. As part of the primary outcome measures, we plan to measure the EGFR expression changes (i.e. EGFR modulation) between buccal smears and bronchial tissues after induction therapy.

SECONDARY OUTCOMES:
Incidence of EGFR mutations | Up to 5 years post-treatment
  The frequency of EGFR mutations in resected tumor specimens following neoadjuvant platinum-based therapy will be evaluated.
Evaluation of immune-based biomarkers | Up to 5 years post-treatment
  The correlation among various continuous and discrete biomarkers will be assessed first by exploratory data analysis using scatter plot matrix, bx plots, BLiP plot, and trellis plots. Correlation among continuous biomarkers will be estimated by Pearson or Spearman rank correlation coefficient. The association on discrete biomarkers will be tested by chi-square or Fisher's exact test. McNamar's test will be applied to test the change of a single discrete biomarker over time.
Time to progression | Up to 5 years post-treatment
  Estimated by Kaplan-Meier method. The Cox (proportional hazards) model will be fitted to estimate the effect of biomarker and other covariates on survival.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cascone, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cascone T, Gold KA, Swisher SG, Liu DD, Fossella FV, Sepesi B, Pataer A, Weissferdt A, Kalhor N, Vaporciyan AA, Hofstetter WL, Wistuba II, Heymach JV, Kim ES, William WN Jr. Induction Cisplatin Docetaxel Followed by Surgery and Erlotinib in Non-Small Cell Lung Cancer. Ann Thorac Surg. 2018 Feb;105(2):418-424. doi: 10.1016/j.athoracsur.2017.08.052. Epub 2017 Dec 6. PMID 29217088
- See also: MD Anderson Cancer Center — http://www.mdanderson.org